CLINICAL TRIAL: NCT06807320
Title: CLINICAL and RADIOGRAPHIC COMPARISON of MINERAL TRIOXIDE AGGREGATE and CALCIUM HYDROXIDE AS INDIRECT PULP CAPPING AGENTS in PRIMARY MOLARS: a RANDOMIZED CLINICAL TRIAL
Brief Title: COMPARISON of MINERAL TRIOXIDE AGGREGATE and CALCIUM HYDROXIDE AS INDIRECT PULP CAPPING AGENTS in PRIMARY MOLARS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, RANA AHMAD, ASSISTANT PROFESSOR, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: F.1-1/2015/ERB/SZABMU/ERB
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Indirect Pulp Cap
Keywords: Indirect Pulp cap; primary molar; MTA
MeSH Terms: interventions — Calcium Hydroxide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group I patients, Calcium hydroxide (Active Comparator): For Group I patients, Calcium hydroxide (Dycal_ Ivory,Dentsply Caulk, Dentsply, L.D. Caulk, Milford, DE,USA ) was used. The catalyst and paste were mixed as per the manufacturer's recommendations.
  Interventions: Drug: Calcium Hydroxide (Ca(OH)2)
- Group II patients, MTA (Experimental): MTA powder ( ProRoot; Dentsply ⁄ Tulsa Dental, Tulsa, OK,USA) was added to sterile water. The mixture was left to achieve a sandy consistency for about thirty seconds. Then, the material was applied to the cavity using a ball condenser.
  Interventions: Drug: MTA pulp dressing material

INTERVENTIONS:
Drug: MTA pulp dressing material — MTA powder ( ProRoot; Dentsply ⁄ Tulsa Dental, Tulsa, OK,USA) was added to sterile water. The mixture was left to achieve a sandy consistency for about thirty seconds. Then, the material was applied to the cavity using a ball condenser.
  Arms: Group II patients, MTA
Drug: Calcium Hydroxide (Ca(OH)2) — For Group I patients, Calcium hydroxide (Dycal_ Ivory,Dentsply Caulk, Dentsply, L.D. Caulk, Milford, DE,USA ) was used. The catalyst and paste were mixed as per the manufacturer's recommendations.
  Arms: Group I patients, Calcium hydroxide

SUMMARY:
The study is designed as randomized clinical trial performed at the Department of Pediatric Dentistry , Pakistan Institute of Medical Sciences (PIMS) , Islamabad on primary molars requiring indirect pulp treatment in patients aged 5 to 9 years. Two groups , I and II of 40 teeth each will be selected according to inclusion criteria . In Group I , indirect pulp capping will be done with Calcium hydroxide while in Group II , it will be done with MTA . Both the groups will be evaluated clinically and radiographically at 0, 3 and 6 months . Results were compiled and analyzed using standard statistical techniques.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Criteria :

  * Primary molars with deep carious lesions
  * No H/O spontaneous pain
  * No associated swelling
  * No tenderness to percussion
  * Absence of pathological mobility
  * No sinus tract
  * Restorable

Radiographic Criteria :

* No periapical radiolucency
* No loss of lamina dura
* No physiological root resorption
* Teeth with radiographic evidence of more than 0.25mm remaining dentin thickness
* No furcal radiolucency

Exclusion Criteria:

* Non restorable teeth

  * Teeth with pathological mobility
  * Teeth with extensive external/internal root resorption.
  * Teeth with pulp canal calcifications
  * Subjects inability to tolerate any of the dental products being used
  * Systemic disease or severe medical complications ; Lack of compliance

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Dentine bridge thickness (DBT) | 3 and 6 months follow up appointment in all successful cases.
  Dentine bridge thickness (DBT) was measured at the 3 and 6 months follow up appointment in all successful cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Pakistan Institute of Medical Sciences, Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided